CLINICAL TRIAL: NCT05183334
Title: Combined On-demand Sildenafil Citrate and Tramadol Hydrochloride for Treatment of Premature Ejaculation: A Randomized Placebo-controlled Double-blind Clinical Trial
Brief Title: Combined On-demand Sildenafil Citrate and Tramadol Hydrochloride for Treatment of Premature Ejaculation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Kamel Abdel Rahman, DR, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: sildenafil and tramadol in PE
Record Dates: First submitted 2021-12-21; First posted 2022-01-10 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Premature Ejaculation
MeSH Terms: conditions — Premature Ejaculation | interventions — Sildenafil Citrate; Tramadol; tamol

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- group 1 (Placebo Comparator): patients with PE
  Interventions: Drug: Placebo
- group2 (Experimental): patients with PE
  Interventions: Drug: Sildenafil 50 mg
- group 3 (Experimental): patients with PE
  Interventions: Drug: Tramadol Hydrochloride 100 MG
- group 4 (Experimental): patients with PE
  Interventions: Drug: Sildenafil 50 mg; Drug: Tramadol Hydrochloride 100 MG

INTERVENTIONS:
Drug: Sildenafil 50 mg — PD5I
  Other Names: sildanafil
  Arms: group 4; group2
Drug: Placebo — placebo
  Other Names: no drug
  Arms: group 1
Drug: Tramadol Hydrochloride 100 MG — opiod
  Other Names: tamol
  Arms: group 3; group 4

SUMMARY:
Premature Ejaculation (PE) is a common sexual dysfunction that has a negative impact on both sex partners. Several lines of treatment have been proposed for the treatment of PE i.e. psychological, behavioral, physiotherapeutic, and pharmacological therapies.Several treatment options have been proposed for treatment of PE including tramadol HCl and PDE5 inhibitors Tramadol HCl is thought to exert its therapeutic action in PE patients

DETAILED DESCRIPTION:
It's clear that PE poses much burden not only on the patient sexual life but also on all aspects of the life of both the patient and his partner. Several treatment options have been proposed for treatment of PE including tramadol HCl and PDE5 inhibitors

. Tramadol HCl is thought to exert its therapeutic action in PE patients through one or more of the following mechanisms: weak µ-opioid effect, 5-HT2 receptor antagonist effect, N-methyl-D-aspartate receptor antagonist effect, serotonin and norepinephrine reuptake inhibitory effect , and acetylcholine receptor antagonist effect . On the other hand, PDE5 inhibitors are thought to play a therapeutic role in treating PE though the following mechanisms: peripheral delay of ejaculation through modulation of contractions of the vas deferens, seminal vesicles, prostate and urethra, increasing the duration of erection , central decrease of the sympathetic output via modulation of NO activity in the medial pre-optic area , peripheral analgesic effect, peripheral analgesic effect, increasing patient confidence, and improving the perception of ejaculation control and sexual satisfaction .

ELIGIBILITY:
Inclusion Criteria:

* no previous medical treatment for PE
* history of premature ejaculation (PE), primary or secondary, and a maximum IELT of 2 minutes prior to treatment.

Exclusion Criteria:

* drug noncompliance, positive history of diabetes mellitus, psychological problems, neurological disorders, erectile dysfunction, chronic illnesses, interpersonal troubles with the spouse, as well as long term medications that could affect the patient condition.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — male act
Enrollment: 160 (Estimated)
Dates: Start 2021-12-30 (Estimated); Primary Completion 2022-12-25 (Estimated); Study Completion 2022-12-25 (Estimated)

PRIMARY OUTCOMES:
satisfaction score | 8week
  sore of sexual satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: ahmed reda, MD, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdel-Hamid IA. Phosphodiesterase 5 inhibitors in rapid ejaculation: potential use and possible mechanisms of action. Drugs. 2004;64(1):13-26. doi: 10.2165/00003495-200464010-00002. PMID 14723556
- [Background] Abu El-Hamd M, Abdelhamed A. Comparison of the clinical efficacy and safety of the on-demand use of paroxetine, dapoxetine, sildenafil and combined dapoxetine with sildenafil in treatment of patients with premature ejaculation: A randomised placebo-controlled clinical trial. Andrologia. 2018 Feb;50(1). doi: 10.1111/and.12829. Epub 2017 May 12. PMID 28497478